CLINICAL TRIAL: NCT04251637
Title: Non Invasive Cardiac Output Evaluation With Starling SV for Lung Elective Surgery
Acronym: NICOLE
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0016; 2019-A01872-55 (Other: ID-RCB)
Record Dates: First submitted 2019-08-01; First posted 2020-02-05 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Thoracic; Surgery
Keywords: esophageal Doppler; thoracic surgery; pulmonary exeresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adult patients scheduled for thoracic pulmonary: Adult patients scheduled in Louis Pradel hospital operating theater (Lyon University Hospital) for elective Lung surgery (lobectomy, bilobectomy or pneumonectomy); by thoracotomy and / or thoracoscopy.
  - Having stated their non opposition to be part of this protocol
  Interventions: Other: Cardiac output monitoring with Starling SV.

INTERVENTIONS:
Other: Cardiac output monitoring with Starling SV. — Intraoperative monitoring of cardiac output by esophageal Doppler, NICOM Starling SV and collection of values for each patient at at least 7 predefined intraoperative times.

SUMMARY:
Intraoperative hemodynamic optimization decreases postoperative complications and length of stay in high risk patient. Therefore, continuous monitoring of cardiac output (Qc) is recommended to guide fluid management. Thoracic bio-reactance is a recent technique that allows cardiac output non-invasive monitoring. However, additional clinical validation studies in humans are required to better define the typologies of patients for whom this monitoring could be proposed routinely. Lung surgery is defined as an intermediate or high risk surgery regarding postoperative cardiac complications. However, surgical patients rarely benefit from continuous monitoring of cardiac output, the available methods being considered too invasive or insufficiently reliable in daily practice. Thoracic bio-reactance (Non Invasive Cardiac Output Monitor (NICOM) Starling SV) has not been studied in this subgroup of clinically relevant patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Scheduled in Louis Pradel hospital operating theater (Lyon University Hospital) for elective Lung surgery (lobectomy, bilobectomy or pneumonectomy); by thoracotomy and / or thoracoscopy.
* Having stated their non opposition to be part of this protocol

Exclusion Criteria:

* Pregnant women ;
* unemancipated minors;
* Persons unable to express their consent;
* Patients with contraindications to the placement of an oesophageal Doppler probe
* Patients with suspicion of pathology or oesogastric lesion (dysphagia, diverticulum, stenosis ...)
* Patients known for stage 2 or higher oesophageal varices
* Patients with a history of significant mediastinal irradiation, or bariatric surgery.
* Patients who have been treated in a therapeutic trial within 30 days of enrollment or who wish to participate in an ongoing study that may interfere with this study.
* Persons benefiting from legal protection measures;
* Patients unable to understand study objectives or refusing to comply with postoperative instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Adult patients scheduled in Louis Pradel hospital operating theater (Lyon University Hospital) for elective Lung surgery (lobectomy, bilobectomy or pneumonectomy); by thoracotomy and / or thoracoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2021-03-13 (Actual); Study Completion 2021-03-13 (Actual)

PRIMARY OUTCOMES:
cardia output measurement | Day 0
  The primary endpoint is the accuracy of the cardiac output value measured with the NICOM Starling SV vs. oesophageal Doppler in thoracic controlled pulmonary exeresis surgery in adults. The accuracy considered valid and reliable will be defined as the error percentage for the Cardiac Output (CO) with an acceptability (concordance) threshold of 30 %. The accuracy will be evaluated on the totality of the time points of interrest.
  All data will be recorded at several time points interest (T0-T7) during surgery:
  * T0 Post Induction / supine position
  * T1 Lateral position closed Thorax / bipulmonary ventilation
  * T2 Lateral position closed Thorax / selective unipulmonary ventilation.
  * T3 Lateral position open Thorax
  * T4 pleural cavity being Washed
  * T5 Before Lung Recruitment Maneuver
  * T6 During Positive End Expiratory Pressure (PEEP) Standardized Pulmonary Recruitment Maneuver 30 cmH20 30 seconds
  * T7 End of Surgery / Awakening in lateral decubitus

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Louis Pradel, Lyon, France

REFERENCES:
- [Derived] Fellahi JL, Abraham P, Tiberghien N, Coelembier C, Maury JM, Bendjelid K. Non-invasive continuous cardiac output monitoring in thoracic cancer surgery: A comparative study between calibrated pulse contour analysis and chest bioreactance. Eur J Anaesthesiol Intensive Care. 2022 Sep 15;1(4):e006. doi: 10.1097/EA9.0000000000000006. eCollection 2022 Aug. PMID 39917369